CLINICAL TRIAL: NCT00003927
Title: High-Dose Infusional Taxol, Amifostine, Doxorubicin, and Cyclophosphamide Followed by Stem Cell Rescue for High Risk Primary and Responsive Metastatic Breast Cancer
Brief Title: Combination Chemotherapy, Amifostine, and Peripheral Stem Cell Transplantation in Treating Patients With Stage II, Stage III, or Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99002; P30CA033572 (NIH); CHNMC-IRB-99002; ALZA-CHNMC-IRB-99002; NCI-G99-1527; CDR0000067115 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-12-11 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Amifostine; Cyclophosphamide; Doxorubicin; Paclitaxel; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- High Dose chemotherapy followed by cell rescue (Experimental): Doxorubicin, cyclophosphamide, Taxol, amifostine
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Amifostine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, amifostine, and peripheral stem cell transplantation in treating patients who have stage II, stage III, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the feasibility of high dose doxorubicin, cyclophosphamide, paclitaxel, and amifostine in patients with high risk stage II/III and responsive stage IV advanced breast cancer. II. Determine the pharmacokinetic profile of paclitaxel administered with amifostine in this regimen in these patients. III. Assess the toxicity of this treatment regimen in this patient population.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously twice daily on days 1-4 for peripheral blood stem cell (PBSC) mobilization and continuing through days 5-10 during PBSC collection. At least 2 weeks following mobilization, patients receive doxorubicin IV as a continuous infusion on days -9 through -5 followed by cyclophosphamide IV over 2 hours on day -5 and amifostine IV over 15 minutes, and paclitaxel IV over 24 hours on day -4. On day -2, 25% PBSC are reinfused and 75% are reinfused on day 0, followed by daily G-CSF subcutaneously or IV beginning on day 1. Patients are followed every 3 months for 2 years, then periodically thereafter.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven breast cancer including: Stage IV metastatic disease with current partial or complete response to prior induction chemotherapy High risk primary disease with less than 60% chance of progression free survival at 3 years Stage II tumors with 10 or more axillary node involvement Stage IIIA or IIIB tumors No bone marrow metastases No CNS metastases No more than 10 bone metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 59 and under Menopausal status: Not specified Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Neutrophil count greater than 2,000/mm3 Platelet count greater than 150,000/mm3 Hemoglobin greater than 9 g/dL (blood transfusions allowed) Hepatic: Bilirubin no greater than 1.2 mg/dL SGOT or SGPT less than 1.5 times upper limit of normal Renal: Creatinine no greater than 1.2 mg/dL Creatinine clearance at least 80 mL/min No prior hemorrhagic cystitis Cardiovascular: Ejection fraction at least 55% by MUGA No prior valvular heart disease or arrhythmia Pulmonary: DLCO at least 60% lower limit of predicted pCO2 no greater than 43 mmHg on room air pO2 greater than 85 mmHg on room air FEV 1 at least 2 liters Other: No other prior malignancy except basal or squamous cell skin cancer, or carcinoma in situ or stage I carcinoma of the cervix Not pregnant HIV negative Hepatitis B negative No prior history of disabling psychosocial disorder No other CNS dysfunction

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No more than 2 prior chemotherapy regimens for metastatic disease Prior total doxorubicin dose no greater than 180 mg/m2 Prior total paclitaxel dose no greater than 750 mg/m2 Endocrine therapy: At least 4 weeks since prior hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy No prior radiotherapy to the left chest wall No prior radiotherapy to greater than 20% of bone marrow (excluding syngeneic transplantation candidates) Surgery: Not specified

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 1999-05-18 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of high dose chemotherapy in advance breast cancer patients. | Up to death

CONTACTS AND LOCATIONS:
Overall Officials: Sayeh Lavasani, MD, Study Chair — City of Hope Medical Center
Locations (1):
- Cancer Center and Beckman Research Institute, City of Hope, Duarte, California, United States